CLINICAL TRIAL: NCT06418555
Title: The Effectiveness of a Digital Home-based Cardiac Rehabilitation Program for TAVR Patients Based: a Randomized Controlled Trial
Brief Title: Construction and Application Plan of Home Cardiac Rehabilitation for Patients Undergoing TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-0921
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-05

CONDITIONS: Aortic Stenosis
Keywords: Cardiac Rehabilitation; Extended Care; Aortic Stenosis; TAVR
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home Rehabilitation Team (Experimental): Adding an immediate information-based intervention to the routine home care intervention with a home cardiac rehabilitation program intervention for TAVR patients.
  Interventions: Behavioral: A home rehabilitation program centered on exercise
- Routine care group (Experimental): Routine care
  Interventions: Behavioral: A home rehabilitation program centered on exercise

INTERVENTIONS:
Behavioral: A home rehabilitation program centered on exercise — Establish a multidisciplinary team, with team members combining clinical experience, summarizing the best evidence as the basis, and using the theory of behavior change wheels as the framework, to preliminarily construct a home-based cardiac rehabilitation plan suitable for TAVR patients in China's national conditions. Conduct expert consultation using the Delphi method to form the final version of the home cardiac rehabilitation plan for TAVR patients.

SUMMARY:
Cardiac rehabilitation is a long-term process, but patients have poor compliance with cardiac rehabilitation. The theory of behavior change rotation aims to comprehensively intervene from three aspects: ability, opportunity, and motivation, promoting individual behavior change by selecting the best intervention function and maximizing the use of available resources. To improve the compliance of TAVR patients with digital home cardiac rehabilitation, this study is based on the needs of TAVR patients and their caregivers for digital home cardiac rehabilitation. Based on the best evidence summary of TAVR patients' home cardiac rehabilitation, a home cardiac rehabilitation plan for TAVR patients is constructed using the theory of behavior change wheels. The Delphi method is used to revise the plan, develop a TAVR patient home cardiac rehabilitation management system, and conduct clinical application research on the plan to explore the intervention effect of TAVR patients' home cardiac rehabilitation based on real-time information intervention.

DETAILED DESCRIPTION:
Conduct home cardiac rehabilitation assessment 1-6 days before discharge; In the first week after discharge, cultivate the patient's motivation for rehabilitation; In the second week after discharge, create a home rehabilitation environment; In the third week after discharge, health education on risk factor management; Health education on anticoagulation management in the fourth week after discharge; 5 weeks after discharge, home symptom and follow-up management education; Carry out home exercise and monitoring from 1 to 12 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing TAVR who were classified as Grade I-III by the New York Heart Association (NYHA); Patients are able to use mobile devices such as smartphones; Patients who have obtained admission qualifications after undergoing digital home cardiac rehabilitation risk assessment by the rehabilitation team; The patient and their family members voluntarily participate in this study and are willing to provide an informed consent form; Able to use remote rehabilitation diagnosis and treatment systems Exclusion Criteria: Malignant tumors or those with serious complications; Patients with hearing and visual impairments; Patients with limited physical activity due to other diseases; Patients with obvious cognitive or mental disorders; Patients without Internet connection after returning home from hospital; Patients who have participated in or participated in other trials or rehabilitation plans within the past three months.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Home-based cardiac rehabilitation exercise adherence | After surgery, and 3 months after discharge
  Measured at the time of the patient's follow-up visit to the clinic

SECONDARY OUTCOMES:
Modified Barthel Index | After surgery, and 3 months after discharge
  Measured at the time of the patient's follow-up visit to the clinic
Minnesota Living with Heart Failure questionnaire | After surgery, and 3 months after discharge
  Measured at the time of the patient's follow-up visit to the clinic
Tilburg Frailty Indicator | After surgery, and 3 months after discharge
  Measured at the time of the patient's follow-up visit to the clinic
Postoperative related complications | After surgery, and 3 months after discharge
  Measured at the time of the patient's follow-up visit to the clinic

CONTACTS AND LOCATIONS:
Overall Officials: Yingying Jia, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Yingying Jia, Zhejiang, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jia YY, Dong MQ, Feng J, Hu JN, Hu HT, Yuan TM, Song JP. The effectiveness of a nurse-led home-based cardiac rehabilitation based on instant information intervention in the prognosis of patients with TAVR: A randomized controlled trial protocol. Curr Probl Cardiol. 2025 Mar;50(3):102967. doi: 10.1016/j.cpcardiol.2024.102967. Epub 2024 Dec 8. PMID 39657845